CLINICAL TRIAL: NCT01261143
Title: Phase III Randomized, Double-blind Study to Assess the Efficacy and Safety of α-lipoic Acid Versus BK-C-0701 in Subjects With Diabetic Neuropathy
Brief Title: Randomized, Double-blind Study to Assess the Efficacy and Safety of α-lipoic Acid Versus BK-C-0701 in Subjects With Diabetic Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Hunjun Jang, bukwang
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BK-C-0701-301
Record Dates: First submitted 2010-12-10; First posted 2010-12-16 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2011-10

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- BK-C-0701, diabetic neuropathy (Experimental)
  Interventions: Drug: BK-C-0701
- alpha lipoic acid, diabetic neuropathy, capsule (Active Comparator)
  Interventions: Drug: BK-C-0701

INTERVENTIONS:
Drug: BK-C-0701 — tablet, 8 weeks

SUMMARY:
The purpose of this study is to determine the:

Primary end point

* change of Total symptom score

Secondary end point

* neurological test

DETAILED DESCRIPTION:
total symptom score shall be calculated from the data of burning, numbness, stabbing pain, paraesthesiae.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus (Type I or II), as defined by the American Diabetes Association, 1997, lasting 1 year and is well-controlled.
* Patient with symmetric sensory-motor Diabetic Neuropathy which is above stage 2
* Result of pin-prick test is 'absent' or 'reduced'
* HbA1C <10%
* Total Symptom Score ≥ 4 points
* At least 1 of the 4 symptoms of the TSS must have occurred continuously over the last 3 months.
* Patient over 19 years of age
* Female who is postmenopausal or is willing to use an effective method of contraception during the study (Effective method=IUD, spermicide with condom, abstinence) or is surgically sterile (underwent a total hysterectomy or bilateral tubal ligation).

Exclusion Criteria:

* Patient who has Proximal asymmetric neuropathy, cranial neuropathies, truncal radiculopathy, diabetic plexopathies, acute or active mononeuropathies (cranial neuropathies, post-herpes neuralgias)
* Patient who has Neuropathy from alcohol, drug (cisplatin, taxol , etcs), malignant cancer or has a medical history of nerve system disease such as Parkinson's disease/ epilepsy/ Multiple sclerosis, etcs.
* Patient who has nerve system disease which can cause sensory loss Myopathy of any cause.
* Peripheral vascular disease severe enough to cause ischemic ulcers or limb ischemia.
* Patients with diabetic proliferating retinopathy requiring immediately therapy and impending blindness.
* Patients with any active neoplastic disease except benign tumor or nonrecurrent malignant tumor for 5 years.
* Patients with clinically significant cardiac, pulmonary, gastrointestinal, haematological, or endocrine disease that may confound interpretation of the study results or prevent the patient from completing the study.
* Patients with atrial fibrillation.
* Patients who have had organ transplants of any kind.
* Patients with significant hepatic or renal disease (AST, ALT or GGT >2 times normal, serum creatinine >1.8 mg/dL (>159 mmol/l) for males or >1.6 mg/dL (>141 mmol/l) for females).
* Patients with a recent history (within last 12 months) of drug or alcohol abuse.
* Use of any investigational drug (participation in a clinical trial) within last 1 month.
* History of severe or anaphylactic reaction to drugs, sulfur or biologic products.
* Recent (within last 3 months) ketoacidosis or hypoglycaemia, necessitating hospital admission.
* Existing foot ulcers.
* Pregnant or lactating females
* History of allergic reaction to the study medication or its excipients.
* Psychiatric, psychological, or behavioural symptoms that would interfere with the patient's ability to participate in the trial.
* Patient who is not suitable to trial by investigator judgment.
* Patient who does not write informed consent prior to start of trial and cannot comply with the trial requirements.
* Antioxidant therapy (vitamins E > 400 IU, C > 200 mg, and beta-Carotene > 30 mg) or pentoxyphylline within last 1 month before start of trial.
* Use of thioctic acid (> 50 mg), evening primrose oil or any other gamma-linolenic acid containing substance within the last 3 months.
* Use of analgesic within >5times of a half-life before administration of investigational medication.
* Use of anticonvulsants(include Pregabalin), antidepressants within 4 weeks before administration of investigational medication.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
TSS | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung soo Ko, Seoul, South Korea